CLINICAL TRIAL: NCT01154582
Title: Nutritional Quality of Egg Proteins and Effect on Satiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Basic Science
Other Study IDs: OVONUTRIAL
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2010-06

CONDITIONS: Physiology; Nutrition
Keywords: ingestive behavior
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Egg (Experimental)
  Interventions: Dietary Supplement: Egg snack
- Cottage cheese (Experimental)
  Interventions: Dietary Supplement: Cottage cheese

INTERVENTIONS:
Dietary Supplement: Egg snack — subject consume 4 cooked whole eggs, providing 380 kcal
  Arms: Egg
Dietary Supplement: Cottage cheese — Subjects consume 200 g of cottage cheese, providing 380 kcal
  Arms: Cottage cheese

SUMMARY:
The project aims to precisely quantify the postprandial amino acid utilization of egg proteins in vivo in humans, and also to assess their satiating power, in relation with nutrient postprandial waves and incretin secretions. For that purpose, 2 independent studies are conducted. The first one is realized using stable isotopes on 8 volunteers ingesting an egg test meal. The second one is a cross over design performed on 30 volunteers to compare the satiating effect of 2 equivalent snacks: whole eggs or cottage cheese.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* BMI between 18 and 25

Exclusion Criteria:

* Allergy to egg or milk protein
* Digestive or metabolic pathology
* Positiveness to HIV, Hepatitis B and C
* Smokers

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2009-02

PRIMARY OUTCOMES:
energy intake at lunch following the snack
Dietary amino acid utilization
  transfer of stables isotopes used as intrinsic markers of egg proteins to metabolic pools

SECONDARY OUTCOMES:
plasma incretin concentrations
  insulin, glucagon, GLP-1, PYY, ghrelin, GIP
postprandial nutrient waves
  plasma glucose, cholesterol, triglyceride, urea
neoglucogenesis
  Endogenous production of glucose and contribution of dietary amino acids

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre de recherche sur volontaires, Bobigny
  - Centre de recherche sur Volontaires, Nantes

REFERENCES:
- [Derived] Fromentin C, Tome D, Nau F, Flet L, Luengo C, Azzout-Marniche D, Sanders P, Fromentin G, Gaudichon C. Dietary proteins contribute little to glucose production, even under optimal gluconeogenic conditions in healthy humans. Diabetes. 2013 May;62(5):1435-42. doi: 10.2337/db12-1208. Epub 2012 Dec 28. PMID 23274906